CLINICAL TRIAL: NCT03189901
Title: Early Management Strategies of Acute Heart Failure for Patients With NSTEMI
Acronym: EMSAHF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLemer2017030
Record Dates: First submitted 2017-06-09; First posted 2017-06-16 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Early Management; Acute Heart Failure; NSTEMI - Non-ST Segment Elevation MI
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular Management (No Intervention): Patients with acute myocardial infarction(AMI) combined with elevated BNP/NT-proBNP level who treated by regular strategy in guideline.
- Regular management+Levosimendan (Experimental): Patients with acute myocardial infarction(AMI) combined with elevated BNP/NT-proBNP level who treated by regular strategy in guideline and levosimendan.
  Interventions: Drug: Regular management+Levosimendan

INTERVENTIONS:
Drug: Regular management+Levosimendan — Patients are treated with regular management recommended in guidelines and levosimendan.
  Arms: Regular management+Levosimendan

SUMMARY:
There are always poor outcomes in patients with acute myocardial infarction(AMI) combined with elevated BNP/NT-proBNP level. An elevated BNP/NT-proBNP level highly indicates acute heart failure(AHF).Levosimendan is recommended in many clinical trials of heart failure and Chinese heart failure guidelines. As a result, the investigators form a hypothesis that when patients with AMI combined with elevated BNP/NT-proBNP level are in conditions before AHF, to use levosimendan may reduces the risk of heart failure and improve the outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with NSTEMI in outpatient service or admitted to hospital;
2. Patients with an elevated NT-proBNP level;
3. Patients sign the informed consent;

Exclusion Criteria:

1. Patients with hypotension(systolic pressure<100mmHg), creatinine clearance rate<30ml/min or be allergic to levosimendan;
2. Patients whose heart function grade of Killip are Level III~IV;
3. Patients suffering from hepatic failure, renal failure or other diseases which may shorten the lifetime to 6 months(for example tumor);
4. Patients with valvular heart diseases influencing haemodynamics, hypertrophic or restricted cardiomyopathy, constrictive pericarditis, severe pulmonary hypertension or myocarditis;
5. Patients with serum potassium level<3.5mmol/L;
6. Pregnant and lactating women;
7. Patients participating in other relevant clinical studies.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood NT-proBNP Level on 3 Days after Random Allocation | Venous blood is collected 3 days after random allocation. Blood NT-proBNP level is tested 1 month.
  To test the blood NT-proBNP level in clinical labs 3 days after random allocation.
Rate of Change from Baseline Blood NT-proBNP Level on 5 Days after Random Allocation | Venous blood is collected at first medical contact and 5 days after random allocation, and blood NT-proBNP level is tested immediately after blood collection.
  To test the blood NT-proBNP level in clinical labs 5 days after random allocation, and compare it with blood NT-proBNP level tested at first medical contact(baseline).

SECONDARY OUTCOMES:
Acute Heart Failure Attack in Hospital | The data is collected during the in hospital period(an average of 2 weeks). Investigators analyse and summary the statistic difference between two groups through study completion.
  To record the number of times of acute heart failure attack in hospital, then analyse the statistic difference between two groups.
Major Adverse Cardiovascular and Cerebrovascular Events in Hospital | The data is collected during the in hospital period(an average of 2 weeks). Investigators analyse and summary the statistic difference between two groups through study completion.
  Major Adverse Cardiovascular Events include all-cause mortality, cardiac death, non-fatal myocardial re-infarction, acute heart failure and stroke when patients are in hospital. Then the investigators analyse the statistic difference between two groups.
Major Adverse Cardiovascular and Cerebrovascular Events on 6 Months | The data is collected on 6 months after patients discharged. Investigators analyse and summary the statistic difference between two groups through study completion.
  Major Adverse Cardiovascular Events include all-cause mortality, cardiac death, non-fatal myocardial re-infarction, rehospitalization because of acute heart failure and stroke on 6 months. Then the investigators analyse the statistic difference between two groups.
Security evaluation of levosimendan | The data is collected during the time when levosimendan is used(an average of 24 hours). Investigators analyse and summary the statistic difference between two groups through study completion.
  Serious adverse reaction such as shock, malignant arrhythmia and so on.
Health Economics Analysis | The data is collected during the in hospital period(an average of 2 weeks). Investigators analyse and summary the statistic difference between two groups through study completion.
  To do health economics analysis using the data including inpatient days, hospitalization costs.
Rate of Patients Whose Plasma NT-proBNP Level Changes at least 30% on 5 Days after Random Allocation | Venous blood is collected at first medical contact and 5 days after random allocation, and blood NT-proBNP level is tested immediately after blood collection.
  To test the blood NT-proBNP level in clinical labs 5 days after random allocation, then calculate the rate of patients whose plasma NT-proBNP level decreased at least 30%(compared with blood NT-proBNP level tested at first medical contact).

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing China-Japan Friendship Hospital, Beijing, Beijng
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Shengli Oilfield Central Hospital, Dongying, Shandog
  - Binzhou People's Hospital, Binzhou, Shandong
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Tai'an Central Hospital, Tai’an, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Yantaishan Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Qilu Hospital of Shandong University (Qingdao), Qingdao